CLINICAL TRIAL: NCT02450565
Title: Translation and Validation of the Traditional Chinese-Cantonese Version of the Self Completed-Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale
Brief Title: Translation of the Self Completed-Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Choi Siu-wai, Postdoctoral Fellow, The University of Hong Kong
Other Study IDs: Neuropathic Pain Translation
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neuropathic Pain; Chronic Pain; Nociceptive Pain
MeSH Terms: conditions — Neuralgia; Chronic Pain; Nociceptive Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Neuropathic pain subjects: The diagnosis of neuropathic pain will be made by pain specialists based on a detailed history, physical examination, investigation results and medical records.
  Interventions: Other: Questionnaire
- Nociceptive pain subjects: The diagnosis of nociceptive pain will be made by pain specialists based on a detailed history, physical examination, investigation results and medical records.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Neuropathic pain, described as 'pain arising as a direct consequence of a lesion or disease on the somatosensory system', affects up to 3-9.8% of the investigators' population, but is often underdiagnosed and undertreated. As treatment is different for patients with neuropathic pain and nociceptive pain, it is important to screen for neuropathic pain. Commonly employed questionnaire-based diagnostic tools in English speaking countries include the Leeds Assessment of Neuropathic Symptoms and Signs pain scale (LANSS) and Neuropathic pain questionnaire (NPQ). Self-completed LANSS is particularly useful as it is not restricted to clinician's examination and can be applied in large-scale research. S-LANSS has been successfully translated, validated and used successfully in Arabic and Turkish, but it has not been utilised in the Chinese population. As verbal translations of the English questionnaires used at the bedside may be prone to errors in interpretation and requires medical practitioners to interpret the questions. Therefore a translation and validation study is essential.

ELIGIBILITY:
Inclusion Criteria:

1. Native Chinese-Cantonese speaker
2. Aged 18 to 80
3. Presence of pain for more than 3 months
4. Able to understand, read and write Traditional Chinese
5. Able to give informed written consent
6. Ability to complete the questionnaire

Exclusion Criteria:

1. Patients who require active pain treatment and / or intervention within 1 week after the initial consultation
2. Voluntary withdrawal from study at any stage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 pain patients will be recruited. One hundred of these patients will be patients suffering from neuropathic pain, and 100 will be patients with nociceptive pain. The diagnosis of neuropathic or nociceptive pain will be made by pain specialists based on a detailed history, physical examination, investigation results and medical records. The pain specialists' diagnosis will be used for distinguishing between nociceptive and neuropathic pain. Demographic information including age, sex, pain diagnosis and duration, education level, co-existing medical problems and employment status will be recorded. The Cantonese S-LANSS will then be administered to patients to be completed without the help of staff.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Questionnaire can successfully identify subjects with neuropathic pain, or nociceptive pain | One year from commencement of study